CLINICAL TRIAL: NCT00041977
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Determine the Effects of Doxycycline Hyclate 20 Mg Tablets [Periostat(R)] Administered Twice Daily for the Treatment of Acne Rosacea
Brief Title: Determine the Effect of Administering Periostat(R) Twice Daily on Patients With Acne Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CollaGenex Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DERM-303
Record Dates: First submitted 2002-07-19; First posted 2002-07-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-11

CONDITIONS: Acne Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

INTERVENTIONS:
Drug: doxycycline hyclate 20 mg twice daily

SUMMARY:
The purpose of this study is to determine whether Periostat(R), Doxycycline Hyclate 20 mg Tablets, taken twice daily is effective in reducing the red and white heads and overall redness associated with rosacea.

ELIGIBILITY:
Inclusion Criteria

* Healthy, post-pubescent male and females > age 18, with rosacea, 10 to 30, [papules and pustules] and < 2 nodules.
* Presence of moderate to severe erythema.
* Presence of telangiectasia.
* Female patients must utilize one of the following methods of birth control throughout the study: IUD, diaphragm, a condom plus the use of a spermicidal gel or foam, oral contraceptives (provided patient has been utilizing this method for at least 4 months prior to baseline and has not changed the brand within this period). Patients may also participate if they are surgically sterilized, in a monogamous relationship with a sterile partner, or sign an agreement that they will abstain from sexual intercourse during the course of a study.
* Patients must sign an informed consent form.
* Negative pregnancy test and non-lactating.

Exclusion Criteria

* The initiation of a hormonal method of contraception within 4 months of baseline; or discontinuation during the course of study; or change in the actual product within 4 months of baseline or during the study.
* The use of topical acne treatments within 2 weeks of baseline.
* The use of systemic antibiotics within 4 weeks of baseline.
* The use of an investigational drug with 90 days of baseline.
* Pregnant women or women of child-bearing potential who are not using an adequate form of birth control as described in Item 4 of the Inclusion Criteria.
* Nursing women.
* Patients with a known hypersensitivity to tetracyclines.
* Patients on clinically significant, concomitant drug therapy (See section below).
* The use of any acne treatment during the course of the study.
* The use of topical steroids 6 weeks prior to baseline and during the study.
* The use of systemic corticosteroids 6 weeks prior to baseline and during the study.
* The use of vasodilators 6 weeks prior to baseline or during the study.
* The use of α-adrenergic receptor-blocking agents 6 weeks prior to baseline and during the study.

Prohibited Medications:

* Chronic use (> 14 days) of sulfa drugs, erythromycin, cephalosporins, and quinolones.
* The use of tetracycline antibiotics is prohibited.
* Use of any acne treatment during the course of the study, including spironolactone.
* Chronic use (> 14 days) of NSAIDs. Chronic use of aspirin at sub-analgesic doses (< 325 mg q.d.) may be used by those patient requiring platelet aggregation inhibitor.
* Penicillin antibiotics should NOT be used during the course of this trial since the bacteriostatic action of doxycycline may interfere with the bactericidal action of penicillins.
* Antacids and vitamins containing aluminum, calcium, or magnesium may impair drug absorption and should be taken at least 1.5 hours before or 3.0 hours after taking study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Florida, Gainesville, Florida
  - University of Miami Medical Center, Miami, Florida
  - Beer and Houck/Florida Dermatology Institute, West Palm Beach, Florida
  - University of Louisville, Louisville, Kentucky
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - David Pariser, MD, Norfolk, Virginia